CLINICAL TRIAL: NCT04017897
Title: The Combination of Anti-PD-1 With Radiotherapy in Previously Untreated Metastatic Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0461
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: The combination of radiotherapy with anti-PD1 (pembrolizumab or nivolumab)

INTERVENTIONS:
Drug: The combination of radiotherapy with anti-PD1 (pembrolizumab or nivolumab) — Subjects with treatment naïve, surgically unresectable metastatic melanoma stages IIIB to IVM1c will be treated with combination of anti-PD1 (pembrolizumab or nivolumab) and radiotherapy.

SUMMARY:
Currently, the first line treatment options for surgically unresectable metastatic melanoma includes anti-PD1 agents such as nivolumab and pembrolizumab. In western countries, UV associated cutaneous melanoma has 30-40% response rates to immune checkpoint inhibitors (ICIs). However, response rates are lower in Asians. The reason for this discrepancy is attributed to the difference in subtypes since most of the Asian patients are mostly subgrouped as acral lentiginous or mucosal types that are unrelated to UV exposures. Thus, there is an unmet need to bolster the effect of ICIs in these patients.

The combination of radiotherapy with ICIs have been demonstrated by several pre-clinical studies. High dose radiation has shown to promote STING pathway which activates dendritic cells needed in priming phase. In addition, low dose radiation may activate macrophage differentiation. These mechanisms in turn may enhance responses to immunotherapy.

In this study, the investigators aim to evaluate the efficacy and tolerability of anti-PD-1 blockade in combination with radiotherapy in surgically unresectable, treatment naive metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject has provided informed consent prior to initiation of any study-specific activities/procedures
* 2. Male or female age > 20 years at the time of informed consent
* 3. Histologically confirmed diagnosis of unresectable stage III or IV melanoma as per AJCC staging system 8th edition
* 4. Subject with no prior systemic treatment
* 5. Eastern Cooperative Oncology Group (ECOG) Performance Status < 1
* 6. Screening labs performed within 7 days of randomization demonstrating adequate hematologic, coagulation, liver, and kidney functions
* 7. Indications for radiotherapy
* 8. BRAF status must be checked, but patient is eligible regardless of BRAF mutations (BRAF V600 wild type or BRAF V600 mutation positive are both eligible)

Exclusion Criteria:

* 1. Ocular melanoma
* 2. Active brain metastasis (stable after 1 month of radiotherapy, gamma knife surgery or surgery)
* 3. Requires palliative radiotherapy
* 4. Previous treatment with chemotherapy, a CTLA-4 or PD-1/PD-L1 antagonist agent, including treatment in adjuvant setting
* 5. Autoimmune disease requiring chronic treatment with systemic corticosteroids or any other immunosuppressive agents 7 days prior to inclusion. (physiologic dose of prednisolone 10mg or equivalent are accepted)
* 6. Concurrent medical disease which would significantly limit full compliance with the study such as, but not limited to the following: heart failure (III, IV as per NYHA classification), renal insufficiency, active infection (requires negative gest for clinically suspected HIV, hepatitis B virus, hepatitis C virus).

If positive results are not indicative of true active or chronic infection, the subject may enter the study after discussion and agreement between the investigator and medical director.

* 7. Has known malignancy that is progressing and requires active treatment
* 8. Has known psychiatric or substance abuse disorders that would interfere with cooperation requirements of the trial
* 9. Lack of availability for clinical follow-up assessments

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 1 year
  assessment of efficacy of anti-PD1 with radiotherapy in terms of overall response rate (ORR)

SECONDARY OUTCOMES:
treatment-related adverse events (TRAE) | 3 years
rate of progression-free survival (PFS) | 1 year
overall survival (OS) | 1 year
disease control rate (DCR) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee J, Chang JS, Roh MR, Jung M, Lee CK, Oh BH, Chung KY, Koom WS, Shin SJ. Clinical Outcomes of Immune Checkpoint Blocker Therapy for Malignant Melanoma in Korean Patients: Potential Clinical Implications for a Combination Strategy Involving Radiotherapy. Cancer Res Treat. 2020 Jul;52(3):730-738. doi: 10.4143/crt.2019.598. Epub 2020 Feb 13. PMID 32054150
- [Derived] Kim HJ, Chang JS, Roh MR, Oh BH, Chung KY, Shin SJ, Koom WS. Effect of Radiotherapy Combined With Pembrolizumab on Local Tumor Control in Mucosal Melanoma Patients. Front Oncol. 2019 Sep 4;9:835. doi: 10.3389/fonc.2019.00835. eCollection 2019. PMID 31552171